CLINICAL TRIAL: NCT06315660
Title: Virtual Reality Cognitive Behavioral Therapy for Anxiety in a Dual Diagnosis Population: A Randomized Clinical Trial Assessing Acceptance, Feasibility, and Preliminary Efficacy
Brief Title: VR Based Therapy to Treat Anxiety in Dual Diagnosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Sct. Hans (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-2021-627
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Dual Diagnosis; Psychosis; Agoraphobia; Social Anxiety Disorder; Substance Use Disorder
MeSH Terms: conditions — Psychotic Disorders; Agoraphobia; Phobia, Social; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The study is a parallel group, investigator initiated, pragmatic, assessor-blinded, 1:1 randomized, clinical feasibility trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: When a participant is randomized to TAU+VR, the senior researcher reveals the allocation to the assigned clinician via secure e-mail. The assigned clinician then schedules the eight therapy sessions with the participant who is thus unblinded to their treatment allocation. If the participant is randomized to TAU, the assigned clinician will inform the participant as soon as possible. The researchers collecting data from the patient and the researchers performing data analysis remain blinded. There are no circumstances wherein unblinding of outcome assessors or data analysists is permissible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU+VR (Experimental)
  Interventions: Behavioral: Cognitive Miljeu Therapy; Behavioral: Virtual Reality based CBT for Anxiety
- TAU (Active Comparator)
  Interventions: Behavioral: Cognitive Miljeu Therapy

INTERVENTIONS:
Behavioral: Cognitive Miljeu Therapy — TAU is an integrated voluntary inpatient treatment based on the principles of CBT, lasting between 12-20 weeks. This treatment includes exercise, close medical monitoring, group-based CBT for SUD, planning with social services, and is called Cognitive Milieu Therapy.
Behavioral: Virtual Reality based CBT for Anxiety — The experimental intervention is a manualized add-on to TAU and comprises eight sessions of 60 minutes over a period of four weeks. Of these eight sessions, six will include 30 minutes of VR-based behavioral experiments targeting agoraphobic and social fear.
  Arms: TAU+VR

SUMMARY:
Dual diagnosis refers to patients with both severe mental illness and substance abuse. Dual diagnosis is therefore a challenging condition to treat, and the group typically represents the most vulnerable individuals in society. Historically, research on dual diagnosis has been underprioritized, and thus, we still do not know enough about how to best assist this vulnerable group.

However, new studies indicate that virtual reality programs can reduce anxiety in patients with psychotic disorders. They achieve this by providing access to a virtual therapist and lifelike environments where patients can challenge their thoughts about the dangers of navigating the world. For both psychotic disorders and substance abuse, we know that anxiety often plays a role in the clinical picture. Therefore, anxiety almost always has an impact on dual diagnosis patients, where it is crucial in maintaining substance abuse and functional impairment. Despite this, anxiety is rarely a focus in existing treatment options, as it is too resource-intensive in addition to an already intensive treatment process.

This study investigates whether the resource barrier can be overcome and whether hospitalized dual diagnosis patients can experience reduced anxiety, fewer relapses, and better outcomes after discharge when their anxiety is treated through partially automated virtual reality therapy.

DETAILED DESCRIPTION:
Introduction - Dual diagnosis (i.e., comorbid psychosis and substance use disorder) is characterized by more severe psychopathology, higher morbidity, less treatment adherence, and smaller treatment gains compared to psychosis alone. Further, there is a clear association between educational status and both prevalence and mortality of psychosis and substance use. Thus, the debilitating symptoms of these disorders propagate social inequality as well as being a substantial societal burden in purely economic terms. Importantly, this burden seems to increase when patients cannot access evidence-based treatment and recent policy changes mean that the amount of dual diagnosis patients in the Danish mental health services will soon more than triple. Improving the accessibility and efficacy of treatment for this vulnerable population is therefore more than ever, a critical unmet need. For this reason, this study aims to investigate the feasibility, efficacy, and acceptability of a partially auto-mated virtual reality (VR) based psychotherapeutic intervention targeting anxiety in dual diagnosis patients. Social avoidance has been theorized to be a highly relevant treatment target in dual diagno-ses populations since it is thought to play a critical role in maintaining symptoms, worsening mood and functional impairment, and deteriorating treatment adherence. Recent studies have found that VR-based cognitive behavioral therapy for psychosis (CBTp) resulted in significant reductions in anxiety and psychotic symptoms, while being safe and acceptable. Studies also show that this treatment can be automated, thus greatly increasing accessibility of treatment. Further, automatiza-tion allows patients to continue treatment even after hospital discharge, potentially maintaining treatment gains for longer. In short, there are several findings which indicate that automated VR-based CBTp is a promising treatment for dual diagnosis and therefore this present trial will be the first in the world to investigate this.

Background - Though CBTp has been shown to be an effective and safe treatment that patients prefer to medication, it is still poorly implemented in many countries. Only 0.07 % of the 5.5 billion DKK that schizophrenia costs Danish society yearly, are related to contacts with a psychologist or psychiatrist, implying that CBTp is also poorly implemented in Denmark. For dual diagnosis patients, prospects of receiving CBTp are further complicated because hospitals offering CBTp often forward patients with comorbid SUD to municipal services. In addition, the evidence supporting psychotherapy for dual diagnosis is still inadequate and the long-term effect of treat-ment remains unclear. This is likely because psychotherapy can be difficult to access for dual diag-nosis patients, being a long-term and complex intervention, which requires a high level of competence from the administering clinician. The lack of high quality clinical research, along with the complexity of the treatment, represent major barriers for implementation. Incorporating the use of VR technology in high quality clinical research may be one way to develop CBTp towards be-coming more accessible, increase long term efficacy and address anxiety symptoms, and easier to implement.

ELIGIBILITY:
Inclusion criteria

* Adult patients (+18 years) admitted to the standard dual diagnosis treatment program in the Mental Health Services of the Capital Region of Denmark.
* Fulfilling diagnostic criteria for a F20-29 disorder and dependence syndrome of either alcohol or drugs in the ICD-10 diagnostic manual.
* Scoring 6 or above on the avoidance subscale and 66 or above on the distress subscale scale of the O-AS. This corresponds to severe levels of avoidance and distress36.

Exclusion criteria

* Incapable of providing informed consent.
* Insufficient knowledge of the Danish and/or English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Oxford Agoraphobic Avoidance Scale | From enrollment to 3 month post treatment (16.9 weeks)
  The Oxford Agoraphobic Avoidance Scale is a psychometrically validated short-form questionnaire designed specifically to assess anxious avoidance and distress in a population with psychosis
Client Satisfaction Questionnaire | From enrollment to post treatment (4 to 8 weeks)
  The Client Satisfaction Questionnaire is an 8-item scale loading to one factor of satisfaction with mental healthcare service.
Systems Useability Scale | From enrollment to post treatment (4 to 8 weeks)
  The System Usability Scale is a standardized questionnaire designed to provide a quick measure of the user's subjective perception of the usability of a computer system. It will be administered to clinical staff after treatment.

SECONDARY OUTCOMES:
Timeline Followback | From enrollment to 3 month post treatment (16.9 weeks)
  • Timeline Follow Back (TLFB) will be used to measure alcohol and drug consumption the last three month at baseline, post-treatment, and follow-up. TLFB is systematic review of consumption every day for a specific period of time, with adequate psychometric qualities.
The Six-item Positive and Negative Symptom Syndrome Scale | From enrollment to 3 month post treatment (16.9 weeks)
  • The Six-item Positive and Negative Symptom Syndrome Scale (PANSS-6) will be used to measure change in psychosis symptom severity between baseline, post-treatment, and follow-up. PANSS-6 is a clinician administered 6-item scale designed to measure positive and negative symptoms in patients with schizophrenia. It has been translated and validated for a Danish population.
The Social Functioning Scale | From enrollment to 3 month post treatment (16.9 weeks)
  The Social Functioning Scale (SFS) will be used to measure changes in social functioning between baseline, post-treatment, and follow-up. The SFS is a widely used measure of impairment in functioning that has been psychometrically validated for populations with psychosis and translated to multiple languages, including Norwegian.
The Questionnaire about the Process of Recovery | From enrollment to 3 month post treatment (16.9 weeks)
  The Questionnaire about the Process of Recovery (QPR) will be used to measure changes in the experience of recovery between baseline, post-treatment, and follow-up. QPR has been translated to several languages, including Swedish, and has acceptable psychometric properties in term of reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Arnfred, phd, Principal Investigator — Mental Health Centre St. Hans